CLINICAL TRIAL: NCT05709145
Title: Written Endoscopist Recommendation to Improve Adherence to Early Repeat Colonoscopy Within 1 Year in Patients With Inadequate Bowel Preparation.
Brief Title: Written Recommendation to Improve Adherence in Poor Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Miguel Angel Pantaleon Sanchez, MD-PhD at Hospital del Mar, Parc de Salut Mar
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Endo-Remind
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Colonic Disease; Adherence, Patient
Keywords: Colonoscopy; Bowel preparation; Quality; Written recommendation
MeSH Terms: conditions — Colonic Diseases; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written recommendation (Experimental): Patients in the intervention group will receive a report of the colonoscopy that will include a written recommendation that the colonoscopy should be repeated within 1 year.
  Interventions: Other: Written recommendation
- Non Written recommendation (No Intervention): Patients in the control group will receive a report of the colonoscopy without a written recommendation that the colonoscopy should be repeated within 1 year.

INTERVENTIONS:
Other: Written recommendation — Patients in the intervention group will receive a report of the colonoscopy that will include a written recommendation that the colonoscopy should be repeated within1 year.
  The colonoscopy report will included that an adequate intestinal cleansing has not been achieved and therefore it is an invalid exploration. Additionally, a written recommendation indicating that the colonoscopy should be repeated within1 year will be included in the colonoscopy report. This recommendation is addressed both to the clinician who requested the colonoscopy and to the patient himself.
  Arms: Written recommendation

SUMMARY:
Our study aims to improve adherence to international clinical guidelines of repeating colonoscopy within 1 year, when bowel cleansing has failed. To this end, we have designed an ambispective study in patients with inadequately prepared colonoscopy. An intervention group to which a precise written recommendation on the need to repeat the colonoscopy in less than 1 year is attached, compared with a control group to which no written recommendations are provided.

The sample size calculation is 171 patients per arm. In addition, we will quantify the percentage of pre-malignant and malignant lesions detected at repeat colonoscopy. We will also analyze factors that may be related to the recommendation or non-recommendation of repeat colonoscopy, as well as the association of variables related to adherence to repeat colonoscopy at an interval of less than 1 year.

Through our study, we intend to demonstrate that a written recommendation, easily applicable and generalizable, has a positive impact on adherence to clinical follow-up guidelines in patients in whom bowel cleansing has failed.

DETAILED DESCRIPTION:
STUDY HYPOTHESIS

In patients with an inadequately prepared colonoscopy, a written recommendation on the need for repeat colonoscopy in less than 1 year improves adherence.

OBJECTIVES

Main objective

- To evaluate adherence to repeat colonoscopy in less than 1 year, after including an accurate written recommendation, versus not including a written recommendation, in patients with a colonoscopy with inadequate preparation.

Secondary objectives

* Determine the detection rate of adenomas, advanced adenomas, serrated lesions, and cancer in the different groups
* To identify risk factors predicting low adherence to repeat colonoscopy.
* To identify variables that influence the gastroenterologist-endoscopist to write down the need to repeat colonoscopy in less than 1 year.

METHODOLOGY

- Ambispective study in patients with inadequately prepared colonoscopy with a prospective inclusion intervention group to which a precise written recommendation on when the colonoscopy should be repeated is attached, compared with a retrospective cohort control group to which no written recommendations are given.

Study population

- Patients with an inadequately prepared colonoscopy for any indication except colorectal cancer screening.

There are 2 population groups according to the recommendations they received:

1. Control group: No-recommendation group.

   Patients to be included in the retrospective cohort will receive a colonoscopy report that includes that the bowel cleansing was inadequate. However, the report will not include that the colonoscopy should be repeated in less than 1 year.
2. Intervention group: When-to-repeat group

Patients in the intervention group will receive a colonoscopy report that includes that the bowel cleansing was inadequate, and in addition the report will include that the colonoscopy should be repeated within 1 year.

Outcome measures

* Adherence to the recommendation will be considered a repeat colonoscopy at an interval of less than 1 year.
* Inadequate preparation will be evaluated according to the Boston Bowel Preparation Scale as less than 2 points in any segment.
* The physician requesting the baseline colonoscopy will be the one who should request the repeat colonoscopy, following the existing written recommendations and in case there are none, based on his clinical judgment.
* To assess the degree of bowel cleansing, we will use the Boston Bowel Preparation Scale (BBPS), which is the most validated of those available. This scale divides the colon into three segments, assigning each segment a score between 0 and 3 points. The overall score of the colon is between 0 and 9 points, with a higher score being understood as a better prepared colon in terms of cleanliness.
* Variables that are potentially related to leaving a written recommendation on the need to repeat and when by the physician-endoscopist will be collected: adenoma detection rate, experience of the endoscopist, full-time vs. partial-time.
* Variables potentially related to low adherence to repeat colonoscopy will be collected such as: patient age, indication for the test, colonoscopy findings (adenomas, advanced adenoma, ADK), physician requesting the examination (gastroenterologist/primary care/other specialists), patient nationality/language barrier, previous non-appearance, previous colonoscopies.
* To facilitate the written recommendation, in all patients with inadequate bowel preparation, a mandatory tab will be created to be filled in the colonoscopy report related to bowel preparation. In case of selecting inadequate cleansing, the recommendation to repeat the colonoscopy in an interval of less than 1 year will be automatically included in the report.

Sample size

Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a two-sided test, 171 subjects are necessary in first group and 171 in the second to find as statistically significant a proportion difference, expected to be of 0.3 in group 1 and 0.45 in group 2. It has been anticipated a drop-out rate of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a colonoscopy with inadequate bowel preparation for any indication except for colorectal cancer screening

Exclusion Criteria:

* Patients with no indication for repeat colonoscopy due to clinical criteria
* Patients with a recommendation to repeat the colonoscopy with a different interval
* Hospitalized patients
* Patients with special reprogramming circuit (colorectal cancer screening, hospitalized patients, complex polypectomies, revision of polypectomies)
* Incomplete examination for other reasons than intestinal cleansing (stenosis, loops, etc...)
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Adherence to repeat colonoscopy | 1 year after index colonoscopy
  Adherence to repeat colonoscopy within1 year in patients with inadequate bowel preparation colonoscopy.

SECONDARY OUTCOMES:
Overall adenoma detection rate | At the moment of colonoscopy
  Ratio of patients with at least one adenoma lesion in the overall colon
Overall serrated lesion detection rate | At the moment of colonoscopy
  Ratio of patients with at least one serrated lesion in the overall colon
Overall cancer detection rate | At the moment of colonoscopy
  Ratio of patients with at least one cancer in the overall colon
Complete colonoscopy rate | At the moment of colonoscopy
  Ratio of successful complete colonoscopies (cecal intubation or in case of previous surgery, ileocolic anastomosis)
Overall advanced adenoma detection rate | At the moment of colonoscopy
  Ratio of patients with at least one advanced adenoma lesion in the overall colon
Boston Bowel Preparation Scale | At the moment of colonoscopy
  Application of the Boston Bowel Preparation Scale to evaluate colonoscopy bowel cleansing

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

REFERENCES:
- [Background] Schreuders E, Sint Nicolaas J, de Jonge V, van Kooten H, Soo I, Sadowski D, Wong C, van Leerdam ME, Kuipers EJ, Veldhuyzen van Zanten SJ. The appropriateness of surveillance colonoscopy intervals after polypectomy. Can J Gastroenterol. 2013 Jan;27(1):33-8. doi: 10.1155/2013/279897. PMID 23378981
- [Background] Atkin W, Wooldrage K, Brenner A, Martin J, Shah U, Perera S, Lucas F, Brown JP, Kralj-Hans I, Greliak P, Pack K, Wood J, Thomson A, Veitch A, Duffy SW, Cross AJ. Adenoma surveillance and colorectal cancer incidence: a retrospective, multicentre, cohort study. Lancet Oncol. 2017 Jun;18(6):823-834. doi: 10.1016/S1470-2045(17)30187-0. Epub 2017 Apr 28. PMID 28457708
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Lieberman DA, Rex DK, Winawer SJ, Giardiello FM, Johnson DA, Levin TR. Guidelines for colonoscopy surveillance after screening and polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2012 Sep;143(3):844-857. doi: 10.1053/j.gastro.2012.06.001. Epub 2012 Jul 3. No abstract available. PMID 22763141
- [Background] Butterly LF, Nadel MR, Anderson JC, Robinson CM, Weiss JE, Lieberman D, Shapiro JA. Impact of Colonoscopy Bowel Preparation Quality on Follow-up Interval Recommendations for Average-risk Patients With Normal Screening Colonoscopies: Data From the New Hampshire Colonoscopy Registry. J Clin Gastroenterol. 2020 Apr;54(4):356-364. doi: 10.1097/MCG.0000000000001115. PMID 30106836
- [Background] Hassan C, Antonelli G, Dumonceau JM, Regula J, Bretthauer M, Chaussade S, Dekker E, Ferlitsch M, Gimeno-Garcia A, Jover R, Kalager M, Pellise M, Pox C, Ricciardiello L, Rutter M, Helsingen LM, Bleijenberg A, Senore C, van Hooft JE, Dinis-Ribeiro M, Quintero E. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 Aug;52(8):687-700. doi: 10.1055/a-1185-3109. Epub 2020 Jun 22. PMID 32572858